CLINICAL TRIAL: NCT01459185
Title: A Feasibility Study of Adjuvant Chemotherapy With Oral Fluoropyrimidine S-1 for Non-small Cell Lung Cancer
Brief Title: A Feasibility Study of Oral Adjuvant Chemotherapy With S-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tomoshi Tsuchiya (Other)
Responsible Party: Sponsor-Investigator, Tomoshi Tsuchiya, Senior Assistant Professor, Nagasaki University
Organization: Nagasaki University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R000007795
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Adjuvant chemotherapy; oral fluoropyrimidine; S-1; Feasibility study; Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1 (Experimental): Single arm of the patients who received complete resection of pathological stage IB, II, or IIIA Non-small cell lung cancer
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — Chemotherapy comprised eight courses (4-week administration, 2-week withdrawal; total 1 year) of S-1 at 80-120 mg/body/day according to body surface area (BSA)
  Other Names: Oral fluoropyrimidine S-1

SUMMARY:
The investigators confirm the feasibility of 1-year administration of oral fluoropyrimidine S-1 as an adjuvant chemotherapy for the patient who received complete resection of non-small cell lung cancer. The investigators presume they can achieve high completion rate with low toxicity.

DETAILED DESCRIPTION:
Chemotherapy comprised eight courses (4-week administration, 2-week withdrawal) of S-1 (FT, gineracil, oteracil potassium; Taiho Pharmaceutical, Tokyo, Japan) at 80-120 mg/body/day according to body surface area (BSA): BSA <1.25 m2, 80 mg/day; BSA >1.25 m2 but <1.5 m2, 100 mg/day; and BSA >1.5 m2, 120 mg/day. S-1 was administered orally, twice daily after meals, starting within 4 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. NSCLC with histological proof.
2. Pathological stage IB, II, or IIIA NSCLC (fifth edition of UICC/AJCC 1997) after complete resection.
3. No prior treatment except for surgery.
4. Sufficient oral intake.
5. Performance status (PS) 0 or 1.
6. Patients also had to have adequate organ function (3500 <leukocytes < 12,000/mm3; thrombocytes, >100,000/mm3; total bilirubin,<1.5 mg/dl; AST and ALT, less than twice the normal limits at each institution; BUN, <25 mg/dl; creatinine, less than the normal limits at each institution; and creatinine clearance (Ccr))

Exclusion Criteria:

1. History of drug hypersensitivity.
2. Contraindication of oral S-1 administration (refer appended paper).
3. Serious surgical or non-surgical complications
4. Active secondary cancer.
5. Watery diarrhea.
6. Pregnant or lactating women.
7. Male who has intention to make pregnant
8. Patient to whom primary doctor judged inadequate to register.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Completion rate | One year

SECONDARY OUTCOMES:
Incidence and grade of adverse reactions | One year

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Nagayasu, MD. PhD., Study Chair — Division of Surgical Oncology, Department of Translational Medical Sciences, Nagasaki University Graduate School of Biomedical Sciences
Locations (1):
- Division of Surgical Oncology, Nagasaki University Graduate School of BIomedical Sciences, Nagasaki, Nagasaki, Japan